CLINICAL TRIAL: NCT03801655
Title: The Effects of a Probiotic on Emotional and Cognitive Processing in Participants Experiencing Low Mood
Brief Title: OxPALM: Oxford Study on Probiotics and Low Mood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R58085/RE003
Record Dates: First submitted 2018-12-04; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Mood; Cognitive Change
MeSH Terms: interventions — Cellulose; Vegetables

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-Kult (Experimental): 4 capsules/day
  Interventions: Dietary Supplement: Bio-Kult
- Placebo (Placebo Comparator): 4 capsules/day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bio-Kult — 4 capsules/day
  Arms: Bio-Kult
Other: Placebo — 4 capsules/day
  Other Names: Cellulose and vegetable capsules
  Arms: Placebo

SUMMARY:
Probiotics are live bacteria which have been suggested to have beneficial effects not only on gut function but also on psychological and cognitive functioning. This study will investigate how a specific probiotic influences emotional and cognitive processing in participants with low mood.

DETAILED DESCRIPTION:
Current antidepressant treatments, which largely target monoamine pathways, are efficacious in treating many aspects of major depression, however it is estimated that more than 30% of depressed patients fail to respond to standard antidepressant medications. Thus, there is a strong clinical need to identify and investigate novel treatment strategies that target different pathways involved in the pathophysiology of mood disorders.

There is now compelling evidence for a link between the enteric microbiota and brain function. The proliferation of the Bifidobacteria and Lactobacilli strains in the large intestine, have anxiolytic and mnemonic effects in both rodents and humans. The intake of these bacteria as live cultures (probiotics) alters the expression of genes integral to neurodevelopment and complex behaviours in rodents. For instance, the oral administration of Bifidobacteria to rats elevated hippocampal brain-derived neurotrophic factor (BDNF), which may underlie some antidepressant actions . At present, only several probiotics have been examined, but it seems likely that of the 40,000 species in the gut, there will be others with psychotropic properties. A multispecies probiotic (Bio-Kult) that contains several species of Bifidobacteria and Lactobacilli is now available and of the 14 types of bacteria packaged into a capsule, 50% have been shown to have psychotropic effects in animals. Dietary supplementation with Bio-Kult therefore, presents as an optimal strategy to test the influence of beneficial gut bacteria on emotional processing and cognition because, the numerous types of bacteria ingested may have a synergistic effect on the brain and so convey a 'stronger' action compared to single species probiotics.

The translation from rodent to human investigations of probiotics has been surprisingly robust, though many more human studies are necessary. In an important early investigation male and female participants consumed either a fermented milk drink containing Lactobacillus casei Shirota or a placebo. At the end of the three-week intervention, there were no overall changes in self-reported affect. However, when only participants whose baseline mood scores fell in the lowest third of the total range were analysed, probiotic supplementation resulted in significantly more participants self-rating as happy rather than depressed, relative to placebo. These results suggest that the emotional benefits of probiotics may be subject to ceiling effects.

Similar effects have been observed in other investigations of mood. For instance, in a recent randomised controlled trial, healthy participants consumed a placebo product or a mixture of several probiotics (Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, and Lactococcus lactis W19 and W58) over a period of four weeks. Relative to placebo, probiotic-treated participants exhibited substantially reduced reactivity to sad mood (assessed by the Leiden Index of Depression Sensitivity Scale), an effect that was specifically attributable to fewer instances of rumination and aggressive cognitions.

In a randomized and double-blind design, healthy volunteers consumed either a mixture of probiotics (Lactobacillus helveticus R0052 and Bifidobacterium longum) or a placebo over 30 days, after which participants completed a range of self-report measures on mood and distress. Participants also collected urine over 24 hours before and after the intervention, enabling cortisol estimations. Relative to placebo, probiotic-treated participants showed significant declines in self-reported negative mood and distress. Parallel to these changes was a decrease in urinary free cortisol, which is suggestive of a potential mechanism underlying the self-reported affective improvements. Interestingly, a follow-up analysis of the individuals with the lowest stress (indexed by cortisol concentrations) showed similar affective benefits to those with higher cortisol concentrations, to some extent contravening the role of ceiling effects in determining probiotic outcomes.

The Bio-Kult probiotic supplement has been selected for use in the present study because it contains the greatest number of bacterial genera and species currently on the market. In preliminary studies in rats, investigators have found that once daily Bio-Kult feeding for 3 weeks reduces circulating corticosterone, a stress hormone that is the corollary of human cortisol. This appears to be consistent with the above human investigation. Thus, taking into consideration its mentioned association with stress and mood, this probiotic supplement provides an interesting tool to investigate effects on cognition and emotional processing, particularly negative affective biases.

Negative affective biases in emotional processing are highly relevant to clinical mood disorders and they are well-recognised in the aetiology and maintenance of depression, such that depressed individuals are more likely to interpret, focus on and remember negative compared to positive emotional cues in self-relevant neuropsychological tasks. Recent theory suggests that over time this positive change in emotional bias contributes to improved mood, and therefore the investigators will study the effect of Bio-Kult on emotional processing in participants experiencing low mood, compared to a placebo.

Participants will be pre-screened using a standardized self-report measure on mood (Patient Health Questionnaire). After filling in the questionnaire, only those who score between 5 and 19 will be recruited into the study. Participants who are deemed non-eligible after filling in this questionnaire will be notified via email (please see enclosed document 'email to non-eligible participants'). The investigators expect to recruit sixty participants aged between 18-55 years, who will be randomised to receive 4 weeks of Bio-Kult or a matched placebo. This design will be made clear to participants.

Emotional and non-emotional cognition tests include computer-based tasks and questionnaires. Sleep function will be measured by actigraphy. The investigators will also be collecting biological data (blood and saliva) to assess cortisol and immune markers. In addition, participants will be asked to complete questionnaires that are relevant to mood, and anxiety, and to fill in a food diary to test for dietary effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing and able to give informed consent for participation in the study.
* Male or female, aged between 18 and 55 years.
* Body mass index (BMI) within the range of 18.5 - 30 kg/m2.
* Sufficiently fluent in English to understand the tasks and instructions.
* Score between 5 and 19 on the Patient Health Questionnaire (PHQ-9).
* Participants not judged to be at risk of suicide or self-harm (as measured using the SCID) and/or in need of immediate treatment to the discretion of the Investigators.

Exclusion Criteria:

* Current history of Axis I psychiatric disorder except for depression or anxiety;
* Current intake (or intention to take) any medication that may affect the outcomes, including medications affecting brain processing, sedation, and motility (examples include antidepressants, anxiolytics, among others);
* Current psychological therapy;
* Major medical disorders (including diseases affecting the human gastrointestinal tract);
* Intake of any other food supplements which, in the opinion of the Investigators, may affect the results;
* Any significant change in diet which, to the discretion of the Investigators, may affect the results;
* Recent participation in another research trial which, to the discretion of the Investigators, may affect the results (for example, using the same / a similar battery of cognitive / emotional tasks in the last 3 months);
* Dyslexia (given the nature of the computer tasks);
* Any other significant finding arising during the screening/selection process which, in the opinion of the Investigators, may influence the participant's ability to take part in the study or the study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Facial Expression Recognition Task | 2 hours
Emotional Categorization Task | 2 hours
Emotional Recall Task | 2 hours
Emotional Recognition Memory Task | 2 hours
Attentional Dot-Probe | 2 hours
Reward Learning Task | 2 hours

SECONDARY OUTCOMES:
Priming Task | 2 hours
Objective sleep | 2 weeks
  Participants will be asked to wear a watch (actigraphy device) for one week at baseline and again during the last week of treatment to measure objective sleep.
Biological measures: cortisol | 4 weeks
  Assays will be conducted to determine levels of cortisol in plasma and saliva. Blood and saliva samples will be collected at pre- and post-intervention sessions. Saliva will also be collected at home by the participants before pre- and post-intervention sessions.
Biological measures: immune markers | 4 weeks
  Assays will be conducted to determine levels of immune markers in plasma. Blood samples will be collected at pre and post-intervention sessions.
Auditory Verbal Learning Task | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Phil Burnet, PhD, Principal Investigator — University of Oxford
Locations (1):
- Warneford Hospital, Oxford, Oxfordshire, United Kingdom